# **PROTOCOL**

# Title:

Intra-rater reliability and agreement between static balance test using Nintendo Wii Balance Board and gait test under dual-task conditions in community-dwelling older adults.

Date: October 27<sup>th</sup> 2020 **Title:** Agreement and intra-rater reliability between static balance test using Nintendo Wii Balance Board and gait test under dual-task conditions in community-dwelling older adults.

Authors: Martin E <sup>1,2</sup>, Jens<sup>1,2</sup>/Gustav<sup>1,2</sup>, Martin J <sup>1</sup>, Stig<sup>1,2</sup>, Jens<sup>1,2</sup>, Gustav<sup>1,2</sup>

#### Affiliations:

- 1. Department of Geriatric Medicine, Aalborg University Hospital, Aalborg, Denmark
- 2. Department of Clinical Medicine, Aalborg University, Aalborg, Denmark

#### **Background:**

Falls are a major concern for healthcare systems globally and for many older adults. To prevent falls, screening for falls risk followed by intervention on relevant risk factors is important[15]. Numerous falls risk factors have been described in the literature [16], and recently, an increasing interest have evolved around the link between mobility and cognition [2, 8]. In continuation hereof, prior studies have demonstrated an association between executive dysfunction, especially when dual-tasking, and falls [8,17]. Thus, a recent consensus statement has recommended testing for the ability to dual-task when walking [2]. However, practical obstacles may be involved when trying to apply this test on older adults. For instance, the dual-task gait test requires space for a walking path, along with the older adult having sufficient dynamic balancing capabilities to walk unassisted. To optimise recruitment of older adults, the possibility to conduct studies in their homes have shown to be important [18, 19]. Notably, a previous study found measuring of static balance, using a Nintendo Wii Balance Board (NWBB) within this setting feasible [20]. This study will examine whether dual tasking using the NWBB static balance test can be considered a suitable alternative to the dual-task gait test.

## **Objectives:**

This study aims to assess agreement between, and 1-week intra-rater reliability of, the dual-task gait test and the NWBB static balance test in community-dwelling older adults (≥65 years).

### Study design:

Cross-sectional study comparing two dual task tests; the NWBB test and the gait test.

#### Methodology:

Participants: We aim to recruit 30 participants aged 65 years or abovethrough convenience sampling at an senior activity centre in the Municipality of Aalborg. Inclusion critiria is age about 65, the ability to stand for 30 seconds without any aid and the ability to walk 8 meters. Exclusion critiria is dementia as this might affect the cognitive results. Activity centres tend to allure seniors with good physique, hence, there is a risk of selection bias using this type of sampling. We will try to minimize this risk by recruiting widely from the activity center and not only from the physical teams, i.e. gymnastics [12].

Setting and data collection: Testing will be performed at the activity centre on the NWBB [21] and the gait test on 8m [5] of hard floor without carpets or obstacles. Data will be registrered in REDCap [22].



Figure 1. Drawing of WBB and gait test settings.

*Procedure*: The participant will attend two test days separated by 14 days. At the initial test day, participants will complete the Orientation Memory Concentration (OMC) test [23] and fill out a questionnaire to inquire baseline characteristics. The questionnaire include the Tilburg Frailty Scale (TFI) [24], Vulnerable Elders Survey 13 (VES- 13)[25], the Short Falls Efficacy Scale International [26] and questions regarding musculoskeletal complications, neurodegenerative diseases or complications, and use of medicines [3] [6] [7] [11]. Afterwards, participants will undergo the testing procedure includingsingle-task cognitive tests, single-task and dual-task gait , and single- and dual-task NWBB tests in a counter-balanced order

The cognitive tests include a supermarket test [27], an arithmetic test [2], and an animal test [2]. Each participant will complete three trials of 30 seconds of each test for a total of nine trials. The single-task gait test includes three trials of eight-meter walking, with the middle six meter being timed. During the single-task NWBB test, participants will be instructed to stand as still as possible for 30 seconds on a WBB for three trials. For the dual-task tests, the participants will perform the gait and NWBB conditions while carring out the before-mentioned cognitive tests simultaneously. Thus, the participants will conduct nine dual-task gait and NWBB tests, respectively. An overview of the testing procedure is provided in Figure 2.

At the second test day, the participants will perform the testing procedure again including the single-task cognitive test, the single- and dual-task gait test, and the single, and dual-task NWBB test. The order of the test will be identical to the order on the initial test day.

| | | | COGNITION | | |
|---|---|---|---|---|---|
| TESTS | | Supermarket test | Arithmetic test | Animal test | No cognitive (singe task) |
| | Cognitive test | 1. Butcher products | 1. 480 – 7 | 1. Birds | |
| | (single task) | 2. Fruits & vegatables | 2. 420 – 7 | 2. On land | |
| | | 3. Dairy products | 3. 450 – 7 | 3. Sea animals | |
| | Gait test | 1. Dairy products | 1. 220 – 7 | 1. On land | 1. Time 1 |
| | (dual + single) | 2. Butcher products | 2. 250 – 7 | 2. Sea animals | 2. Time 2 |
| | | 3. Fruits & vegatables | 3. 280 – 7 | 3. Birds | 3. Time 3 |
| | WBB test | 1. Fruits & vegatables | 1. 350 – 7 | 1. Sea animals | 1. Area + speed 1 |
| | (dual + single) | 2. Butcher products | 2. 320 – 7 | 2. On land | 2. Area + speed 2 |
| | | 3. Dairy products | 3. 380 – 7 | 3. Birds | 3. Area + speed 3 |

Figure 2. Schematic overview of this study's tests.

Analysis: Data will be used for calculating the correlation between the gait test and the NWBB test using correct response rate (CRR) [8], dual task gait/balance cost (DTGC) and dual task cognition cost (DTCC) [7]. Agreement will be investigated through Bland-Altman plots [13] along with calculation of mean difference, paired t-test, and LOA. Correlation will be shown using Pearson's correlation. Analysis of intra-rater reliability will include interclass coefficient (ICC), coefficient variant (CV), limits of agreement (LOA), standard error of measurements (SEM) and mean difference including paired T-test.

Safety considerations: Participants will be followed closely through the gait test and the NWBB test. If participants are unable to walk 12x8m or unable to keep their balance for 12x30sec the investigator will interrupt the testing and they will be excluded from the study for safety reasons. Smaller breaks and single fails are accepted.

*Reproducibility*: The study is easily reproducible. Participants represents a wider part of the background population between elders above 65yo. Testing only includes a WBB and 8m of firm flat floor without obstacles.

*Ethics*: Participants will participate voluntarily with oral and written consent. The local ethics committee will have consulted, and the study will be registered at the Danish Data Protection Agency.

# Time schedule:

Testing will be conducted throughout November 2020, and the study result will be presented as an article in 2021.

#### Funding:

This study is funded by the Department of Geriatric Medicine, Aalborg University Hospital, Aalborg, Denmark.

#### Conflict of interests:

Investigators in this project has no economical or any other partial interests. One of the employees in the research team at the geriatric department is a co-owner of the software Fysiometer, which is used for data collecting from the WBB, however, he will not participate in any of the data collection or subsequent analyses.

#### References:

- 1. Clark RA, Bryant AL, Pua Y, McCrory P, Bennell K, Hunt M. Validity and reliability of the Nintendo Wii Balance Board for assessment of standing balance. Gait Posture. 2010 Mar;31(3):307–10.
- 2. Cullen S, Montero-Odasso M, Bherer L, Almeida Q, Fraser S, Muir-Hunter S, et al. Guidelines for gait assessments in the canadian consortium on neurodegeneration in aging (CCNA). Can Geriatr J. 2018;21(2):157–65.
- 3. Gobbens RJJ, Boersma P, Uchmanowicz I, Santiago LM. The Tilburg Frailty Indicator (TFI): New Evidence for Its Validity. Clin Interv Aging [Internet]. 2020 Feb 21 [cited 2020 Oct 28]; Volume 15:265–74. Available from: https://www.dovepress.com/the-tilburg-frailty-indicator-tfi-new-evidence-for-its-validity-peer-reviewed-article-CIA
- 4. Gonzalez Da Silva C, Petersson KM, Faísca L, Ingvar M, Reis A. The effects of literacy and education on the quantitative and qualitative aspects of semantic verbal fluency. J Clin Exp Neuropsychol. 2004;26(2):266–77.
- 5. Hunter SW, Divine A, Omana H, Wittich W, Hill KD, Johnson AM, et al. Effect of Learning to Use a Mobility Aid on Gait and Cognitive Demands in People with Mild to Moderate Alzheimer's Disease: Part II-4-Wheeled Walker. J Alzheimer's Dis. 2019;71(s1):S115–24.
- 6. Lamb SE, Jørstad-Stein EC, Hauer K, Becker C. Development of a common outcome data set for fall injury prevention trials: The Prevention of Falls Network Europe consensus. J Am Geriatr Soc. 2005;53(9):1618–22.
- 7. Montero-Odasso M, Almeida QJ, Bherer L, Burhan AM, Camicioli R, Doyon J, et al. Consensus on shared measures of mobility and cognition: From the Canadian Consortium on Neurodegeneration in Aging (CCNA). Journals Gerontol Ser A Biol Sci Med Sci. 2019;74(6):897–909.
- 8. Muir-Hunter SW, Wittwer JE. Dual-task testing to predict falls in community-dwelling older adults: A systematic review. Physiother (United Kingdom) [Internet]. 2016;102(1):29–40. Available from: http://dx.doi.org/10.1016/j.physio.2015.04.011
- 9. Nielsen TR, Waldemar G. Effects of literacy on semantic verbal fluency in an immigrant population. Aging, Neuropsychol Cogn. 2016;23(5):578–90.
- 10. Pellecchia GL. Postural sway increases with attentional demands of concurrent cognitive task. Gait Posture. 2003;18(1):29–34.
- 11. Riis J, Eika F, Blomkvist AW, Rahbek MT, Eikhof KD, Hansen MD, et al. Lifespan data on postural balance in multiple standing positions. Gait Posture [Internet]. 2020;76(October 2019):68–73. Available from: https://doi.org/10.1016/j.gaitpost.2019.11.004
- 12. Witham MD, Stott DJ. Conducting and reporting trials for older people. Age Ageing. 2017;46(6):889–94.
- 13. Martin Bland J, Altman DG. STATISTICAL METHODS FOR ASSESSING AGREEMENT BETWEEN TWO METHODS OF CLINICAL MEASUREMENT. Lancet. 1986 Feb 8:327(8476):307–10.
- 14. Shrout PE, Fleiss JL. Intraclass correlations: Uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420–8.

- 15. Panel on Prevention of Falls in Older People American Geriatrics Society and British Geriatrics Society. Summary of the updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011;59(1):148–57.
- 16. Deandrea S, Lucenteforte E, Bravi F, Foschi R, La Vecchia C, Negri E. Risk factors for falls in community-dwelling older people: a systematic review and meta-analysis. Epidemiology. 2010;21(5):658–68.
- 17. Hsu CL, Nagamatsu LS, Davis JC, Liu-Ambrose T. Examining the relationship between specific cognitive processes and falls risk in older adults: a systematic review. Osteoporos Int. 2012 Oct;23(10):2409-24. doi: 10.1007/s00198-012-1992-z. Epub 2012 May 26. PMID: 22638707; PMCID: PMC4476839.
- 18. Bowsher J, Bramlett M, Burnside IM, Gueldner SH. Methodological considerations in the study of frail elderly people. J Adv Nurs. 1993 Jun;18(6):873-9. doi: 10.1046/j.1365-2648.1993.18060873.x. PMID: 8320380.
- 19. Davies K, Collerton JC, Jagger C, Bond J, Ah Barker S, Edwards J, et al. Engaging the oldest old in research: lessons from the Newcastle 85+ study. BMC Geriatr. 2010 Sep;10(1):64.
- 20. Gustav V. Sørensen, Martin G. Jørgensen, Jesper Ryg, Tahir Masud & Stig Andersen | Selena Gray (Reviewing editor) (2019) Development, feasibility, acceptability, and adjustment of a portable, multifactorial falls risk test battery for community-dwelling older adults., Cogent Medicine, 6:1, DOI: 10.1080/2331205X.2019.1674099
- 21. Jørgensen MG, Laessoe U, Hendriksen C, Nielsen OB, Aagaard P. Intrarater reproducibility and validity of Nintendo Wii balance testing in community-dwelling older adults. J Aging Phys Act. 2014 Apr;22(2):269-75. doi: 10.1123/japa.2012-0310. Epub 2013 May 22. PMID: 23752090.
- 22. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)-A metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009; 42: 377–381.
- 23. Wade DT, Vergis E. The Short Orientation-Memory-Concentration Test: a study of its reliability and validity. Clin Rehabil. 1999 Apr;13(2):164-70. doi: 10.1191/026921599673848768. PMID: 10348397.
- 24. Andreasen J, Sørensen EE, Gobbens RJ, Lund H, Aadahl M. Danish version of the Tilburg Frailty Indicator--translation, cross-cultural adaption and validity pretest by cognitive interviewing. Arch Gerontol Geriatr. 2014 Jul-Aug;59(1):32-8. doi: 10.1016/j.archger.2014.02.007. Epub 2014 Feb 28. PMID: 24680192.
- 25. Saliba D, Elliott M, Rubenstein LZ, Solomon DH, Young RT, Kamberg CJ, Roth C, MacLean CH, Shekelle PG, Sloss EM, Wenger NS. The Vulnerable Elders Survey: a tool for identifying vulnerable older people in the community. J Am Geriatr Soc. 2001 Dec;49(12):1691-9. doi: 10.1046/j.1532-5415.2001.49281.x. PMID: 11844005.
- 26. Kempen, G. I. J. M., Yardley, L., Van Haastregt, J. C. M., Zijlstra, G. A. R., Beyer, N., Hauer, K., & Todd, C. (2008). The short FES-I: A shortened version of the falls effi- cacy scale-international to assess fear of falling. Age and Ageing, 37(1), 45–50. doi:10.1093/ageing/afm157
- 27. Nielsen TR, Waldemar G. Effects of literacy on semantic verbal fluency in an immigrant population. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2016 Sep;23(5):578-90. doi: 10.1080/13825585.2015.1132668. Epub 2016 Jan 20. PMID: 26786839.